CLINICAL TRIAL: NCT05489276
Title: Phase I Clinical Trial of TQB2825 Injection in Subjects With CD20 Positive Hematological Tumors
Brief Title: Clinical Trial of TQB2825 in Subjects With CD20 Positive Hematological Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2825- I-01
Record Dates: First submitted 2022-06-17; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Hematological Tumors
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2825 injection (Experimental): TQB2825 injection is given intravenously every 2 weeks, and every 4 weeks (28 days) as a treatment cycle, with the longest treatment duration not exceeding 2 years.
  Interventions: Drug: TQB2825 injection

INTERVENTIONS:
Drug: TQB2825 injection — TQB2825 injection is a bi-specific, humanized antibody against CD3×CD20, with the structure ratio of anti-CD3 to anti-CD20 of 1:2. It has two asymmetric Fab ends and a complete Fc end, and is a natural IgG4 subtype with weak antibody-dependent cell-mediated cytotoxicity or complement dependent cytotoxicityfunction. By bridging CD3 and CD20, TQB2825 injection induces T cell activation to promote T cell proliferation/expansion, promote the formation of cytolytic synapses, and cause cytotoxic T cells to release perforin and granase, thereby killing CD20 positive tumor cells. Therefore, TQB2825 injection is intended for the treatment of CD20 positive hematologic tumors, including but not limited to lymphoma, leukemia and myeloma.

SUMMARY:
This is a single-group, open, dose escalation and expansion Phase I clinical study, with phase I being a dose escalation study and Phase II being a dose expansion study. The purpose of this study was to evaluate the safety and tolerability of TQB2825 injection in CD20-positive hematological tumor subjects, and to determine dose-limiting toxicity (DLT), maximum tolerated dose (MTD) (if any), or optimal biological dose (OBD), and recommended phase II dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

* 1 Malignant hematologic tumors, including but not limited to lymphoma, leukemia, myeloma, etc., which are clearly diagnosed by histology or cytology (report of immunotyping results is required).
* 2 Immunophenotypic analysis showed CD20 positive.
* 3 18 years old ≤ Age ≤75 years old; Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1; Life expectancy ≥ 3 months.
* 4 Prior induction or salvage therapy ≥second-line treatment, adequate treatment with at least one regimen containing an anti-CD20 mab (combination chemotherapy or monotherapy), and meeting the following criteria:

  1. Patients who have not been alleviated after the last adequate treatment or whose disease has progressed after remission, or who have relapsed after autologous hematopoietic stem cell transplantation (auto-HSCT)
  2. Patients with refractory Anti-CD20 monoclonal antibody.
* 5 According to the 2014 Lugano criteria, there is at least one measurable lesion, that is, a lymph node lesion with a diameter >15 mm or an extranodal lesion with a diameter >10 mm according to the cross-sectional CT image (for tumors with the 2014 Lugano evaluation criteria).
* 6 Negative serum/urine pregnancy test within 7 days prior to initial dosing and must be non-lactating subjects; Female subjects of reproductive age agree to use contraception (such as an intrauterine device, birth control pill, or condom) during the study period and for six months after the study ends; Male subjects agreed to use contraception during the study period and for six months after the end of the study period.
* 7 The subjects voluntarily joined the study and signed informed consent with good compliance.

Exclusion Criteria:

* 1 Tumor diseases and medical history:

  1. Hematologic malignancies that have or are suspected to involve the central nervous system (CNS) or primary CNS lymphoma;
  2. Subjects who had or currently had other malignancies within 3 years. Two conditions can be included in clinical trials: five consecutive years of disease-free survival (DFS) for other malignancies treated with a single operation; Cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor infiltrating basal membrane)];
  3. Clinically significant uncontrolled pleural effusion ascites requiring repeated drainage and pericardial effusion with medium or higher volume.
* 2 Previous anti-tumor therapy:

  1. Prior treatment with other antibodies targeting both CD3 and CD20;
  2. Received any investigational antibody drug therapy, CAR T therapy, or other immunocytotherapy, or auto-HSCT within 3 months prior to initial administration;
  3. Prior allogeneic hematopoietic stem cell transplantation (ALLO-HSCT);
  4. Any major surgery, chemotherapy and/or radiotherapy, immunotherapy or targeted therapy within 4 weeks prior to initial administration;
  5. The half-life of the first administration is less than 5 drugs from the previous oral targeted therapy (calculated from the end time of the last treatment);
  6. Received proprietary Chinese medicines with anticancer indications specified in NMPA approved drug instructions within 2 weeks prior to initial administration;
  7. The toxicity of previous antitumor treatment is not recovered to ≤ grade 1(common terminology criteria for adverse events 5.0) .
* 3 Associated diseases and medical history:

  1. Liver abnormalities: decompensated cirrhosis and active hepatitis;
  2. Renal abnormalities:

     I. Renal failure requiring hemodialysis or peritoneal dialysis; II. Previous history of nephrotic syndrome.
  3. Gastrointestinal abnormalities:

     I. Chronic diarrhea persists despite maximum medical treatment; II. Presence of active inflammatory bowel disease within 4 weeks prior to initial administration.
  4. Cardiovascular and cerebrovascular abnormalities:

     I. With or prior history of central nervous system diseases; II. MRI evidence of brain inflammation and/or vasculitis; III. Occurrence of cerebrovascular accident or cerebral infarction within 6 months before the first administration; IV. Arteriovenous thrombosis events such as deep vein thrombosis and pulmonary embolism occurred within 3 months before the first administration; V. With or prior history of cardiovascular disease; VI. Hypertension that cannot be controlled by the combination of the two drugs (systolic blood pressure ≥160 mmHg and diastolic blood pressure ≥100 mmHg measured at least twice); VII. Previous or current heart valvulitis or endocarditis.
  5. Medical history of immunodeficiency: known human immunodeficiency virus (HIV) infection, or other acquired, congenital immunodeficiency disease;
  6. Uncontrollable systemic bacterial, fungal or viral infection.
  7. Lung disease:

     I. Previous or present with or suspected chronic obstructive pulmonary disease (COPD) and forced expiratory volume at the end of 1 second (FEV1) <60% (estimated value); II. Past or present non-infectious pneumonia requiring corticosteroid treatment; IV. Active tuberculosis.
  8. History of severe allergies of unknown cause; Known allergy to monoclonal antibodies or to exogenous human immunoglobulin; Known allergy to investigational drug excipients.
* 4 Getting a live-attenuated vaccine within 4 weeks prior to initial administration or during planned study period.
* 5 Participated in clinical trials of other drugs within 30 days.
* 6 It is estimated that the compliance of patients participating in this clinical study is insufficient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity（DLT） | 104 weeks
  To evaluate DLT of TQB2825 injection in Chinese adult patients with CD20 positive hematological tumors.
the maximum tolerated dose (MTD) | 104 weeks
  To evaluate MTD of TQB2825 injection in Chinese adult patients with CD20 positive hematological tumors.
Recommended Phase II Dose（RP2D) | 104 weeks
  To evaluate RP2D of TQB2825 injection in Chinese adult patients with CD20 positive hematological tumors.

SECONDARY OUTCOMES:
Adverse events (AE) | Baseline up to 104 weeks
  The occurrence of all adverse events (AE)
serious adverse events (SAE) | Baseline up to 104 weeks
  serious adverse events (SAE)
treatment-related adverse events(TRAE) | Baseline up to 104 weeks
  treatment-related adverse events(TRAE)
Elimination half-life (to be used in one-or non- compartmental model) （t1/2) | Assessments were performed at fixed time points from Cycle 1 to Cycle 6, with each period being 28 days, about 6 months
  t1/2 is time that takes for the blood concentration of TQB2825 or metabolite(s) to drop by half.
Tmax | Assessments were performed at fixed time points from Cycle 1 to Cycle 6, with each period being 28 days, about 6 months
  Time to reach maximum (peak) plasma concentration following drug administration（Tmax)
Maximum (peak) plasma drug concentration （Cmax) | Assessments were performed at fixed time points from Cycle 1 to Cycle 6, with each period being 28 days, about 6 months
  Cmax is the maximum plasma concentration of TQB2825.
Area under the plasma concentration-time curve from time zero to time t （AUC0-t) | Assessments were performed at fixed time points from Cycle 1 to Cycle 6, with each period being 28 days, about 6 months
  To characterize the pharmacokinetics of TQB2825 by assessment of area under the plasma concentration time curve from the first dose to the last measurable concentration point.
Area under the plasma concentration-time curve from time zero to time ∞（AUC0-∞) | Assessments were performed at fixed time points from Cycle 1 to Cycle 6, with each period being 28 days, about 6 months
  To characterize the pharmacokinetics of TQB2825 by assessment of area under the plasma concentration time curve from the first dose to infinity.
Minimum steady-state plasma drug concentration during a dosage interval （Cmin,ss) | Assessments were performed at fixed time points from Cycle 1 to Cycle 6, with each period being 28 days, about 6 months
  Cmin is the minimum plasma concentration of TQB2825
Progress Free Survival（PFS) | up to 96 weeks
  Time from the first dose to the first documentation of PD or death from any cause, whichever occurs first
Disease control rate（DCR) | up to 96 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of Response (DOR) | up to 96 weeks
  The time when the participants first achieved complete or partial remission to disease progression.
Overall survival (OS) | up to 96 weeks
  the time from start of study treatment to date of death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China